CLINICAL TRIAL: NCT01298921
Title: A Pilot Study of Demand Valve Oxygen Inhalation Therapy for Cluster Headache
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left Geisinger-study terminated prematurely - 4 patients enrolled
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0205
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-04

CONDITIONS: Cluster Headache
Keywords: Headache; Cluster Headache; Oxygen Therapy
MeSH Terms: conditions — Cluster Headache; Headache | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continous Flow Oxygen (Active Comparator)
  Interventions: Drug: Oxygen
- Oxygen Demand Valve (Experimental)
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — A demand valve delivers oxygen to the user as soon as they try to inhale from an attached mask or mouth tube. As the user starts to inhale, the slight drop in pressure within the mouth piece or mask lifts a valve and starts the oxygen flow. If the user inhales more deeply, more oxygen will flow in response to the increased demand, hence the name demand valve. Unlike a constant flow O2 regulator, a demand valve has no flow meter or flow rate controls, but it is capable of delivering O2 from 0 to 160 liters per minute (LPM). When using a demand valve, O2 dosage is controlled by respiration rate
  Arms: Oxygen Demand Valve
Drug: Oxygen — 100 percent continuous oxygen given via a non-rebreather facemask at 7 to 15 liters per minute for 20 minutes
  Arms: Continous Flow Oxygen

SUMMARY:
Cluster headache is a disorder marked by frequent attacks of short-lasting, severe, unilateral head pain with associated autonomic symptoms. It is the most severe head pain syndrome known. Currently, the two most common treatments for cluster headaches are inhaled oxygen and injectable sumatriptan. These treatments do not work for all cluster headache patients, and patients who smoke may eventually develop contraindication to triptans. New treatment options are needed.

An alternative method of oxygen delivery (as opposed to continuous flow) uses a demand valve that is controlled by respiration rate, allowing increased oxygen flow in response to increased demand. This system may be more efficacious at stopping a cluster headache attack than the currently prescribed oxygen delivery system.

This study will compare the effectiveness of oxygen delivered via demand valve versus continuous high flow oxygen via non-rebreather face mask in the acute treatment of a cluster headache attack. All patients will treat one cluster headache with each of the 2 treatment methods.

DETAILED DESCRIPTION:
Cluster headache is a primary headache disorder marked by frequent attacks of short-lasting, severe, unilateral head pain with associated autonomic symptoms. The goal of acute therapy for cluster headache is fast, effective and consistent relief.

In the currently recommended dosing strategy of continuous flow 100% oxygen given via a non-rebreather face mask at 7-15L/min, the time to improvement can sometimes take upwards of 20-30 minutes and is not effective for all cluster headache sufferers.

An alternative method of oxygen delivery (versus continuous flow) uses a demand valve which is controlled by the respiration rate, allowing increased oxygen flow in response to increased demand. This delivery system may be better at stopping a cluster headache attack than the continuous flow model as it can support hyperventilation which can enhance cerebral arterial vasoconstriction via a state of hyperoxia and hypocapnia. Arterial vasoconstriction is one hypothesized method by which oxygen can abort a cluster headache attack.

This proof of concept trial will evaluate if oxygen delivered via demand valve with a specific breathing technique is effective as a cluster headache acute treatment and is more effective than the traditional continuous high flow oxygen treatment with a non-rebreather face mask.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 65 with history of moderate severe or very severe cluster headaches and currently in a cluster headache period or cycle are included.

Exclusion Criteria:

* Subjects who have a history of chronic obstructive lung disease, those who have major neurologic disorders other than cluster headaches, those with a history of syncope, or lightheadedness with hyperventilation and pregnant women are excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd D. Rozen, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania, United States

REFERENCES:
- [Derived] Rozen TD, Fishman RS. Demand valve oxygen: a promising new oxygen delivery system for the acute treatment of cluster headache. Pain Med. 2013 Apr;14(4):455-9. doi: 10.1111/pme.12055. Epub 2013 Jan 31. PMID 23369112
- See also: Geisinger Health System — http://www.geisinger.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the enrollment of 4 participants in this study, the PI left Geisinger and the study was terminated. Geisinger does not have any details regarding which Arm/Group participants completed. Therefore, 0 was added as the enrollment for each group.
Groups:
- Continous Flow Oxygen: Oxygen : 100 percent continuous oxygen given via a non-rebreather facemask at 7 to 15 liters per minute for 20 minutes
- Oxygen Demand Valve: Oxygen : A demand valve delivers oxygen to the user as soon as they try to inhale from an attached mask or mouth tube. As the user starts to inhale, the slight drop in pressure within the mouth piece or mask lifts a valve and starts the oxygen flow. If the user inhales more deeply, more oxygen will flow in response to the increased demand, hence the name demand valve. Unlike a constant flow O2 regulator, a demand valve has no flow meter or flow rate controls, but it is capable of delivering O2 from 0 to 160 liters per minute (LPM). When using a demand valve, O2 dosage is controlled by respiration rate
Period: Overall Study
Arm/Group | Continous Flow Oxygen | Oxygen Demand Valve
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: After the enrollment of 4 participants in this study, the PI left Geisinger. Geisinger does not have any details regarding which Arm/Group participants completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Continous Flow Oxygen | Oxygen Demand Valve | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical — After the enrollment of 4 participants in this study, the PI left Geisinger. Geisinger does not have any details regarding which Arm/Group participants were assigned to.
Sex: Female, Male — After the enrollment of 4 participants in this study, the PI left Geisinger. Geisinger does not have any details regarding which Arm/Group participants were assigned to.
Count of Participants — After the enrollment of 4 participants in this study, the PI left Geisinger. Geisinger does not have any details regarding which Arm/Group participants were assigned to.

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Headache Pain
Description: Headache response after 30 minutes of oxygen treatment. Headache response is defined as a reduction in headache pain intensity from moderate, severe, or very severe pain to mild or no pain.
Time Frame: 30 minutes
Population: Data cannot be found despite efforts to contact primary investigator. Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data for pre-specified Primary and Secondary Outcome Measures to report in Outcome Measure data table(s).
Arm/Group | Continous Flow Oxygen | Oxygen Demand Valve
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Headache Relief and Pain Free
Description: 1. Percentage of patients with no pain after 30 minutes of treatment
  2. Headache relief and pain free at other time points (5 to 60 minutes)
  3. Reduction of autonomic symptoms at 30 minutes
  4. Any difference in treatment response between episodic and chronic cluster headache patients (if patient #'s allow)
  5. Rescue medication use
  6. Cluster headache recurrence by 24 hours post oxygen treatments
  7. Patient satisfaction with treatment response compared with prior oxygen treatment if have utilized8.Likelihood of choosing this technique again to treat a cluster headache attack
Time Frame: 5 to 60 minutes
Population: as for outcome 1
Arm/Group | Continous Flow Oxygen | Oxygen Demand Valve
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Data cannot be found despite efforts to contact primary investigator. Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data for pre-specified Primary and Secondary Outcome Measures to report in Outcome Measure data table(s).
Arm/Group | Continous Flow Oxygen | Oxygen Demand Valve
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No